CLINICAL TRIAL: NCT01577407
Title: Non Opioid Treatment for Experimental Dyspnea
Acronym: Nefopel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P 110103
Record Dates: First submitted 2012-02-23; First posted 2012-04-13 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2011-10

CONDITIONS: Dyspnea; Pain
Keywords: Dyspnea; Pain
MeSH Terms: conditions — Dyspnea; Pain | interventions — Nefopam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nefopam (Experimental)
  Interventions: Drug: Nefopam
- placebo (Placebo Comparator)
  Interventions: Drug: Nefopam

INTERVENTIONS:
Drug: Nefopam — Subjects will be infused intravenously with nefopam (20mg/2mL) over a course of 30 minutes in a supine position. There will be a single administration of IV 20 mg nefopam and IV placebo. Each intervention will occur on a separate day.
  Other Names: acupan

SUMMARY:
The purpose of this protocol is to test the effects of the non opioid nefopam on experimental dyspnea and on the counterirritation (ie inhibition of one pain by another pain) induced by dyspnea in healthy subjects.

DETAILED DESCRIPTION:
Dyspnea and pain share many features. One of them is the counterirritation phenomenon: defined in pain research as the attenuation of one pain by another pain. Dyspnea induced with inspiratory threshold loading (increased sense of work/effort ) has been shown to attenuate electrical pain as shown through nociceptive flexion reflex inhibition, or thermal pain, as measured with cortical evoked responses (laser evoked potentials-LEP).

The investigators will study whether nefopam modulates the counterirritation of laboratory induced dyspnea in healthy subjects. The effect of nefopam on experimental dyspnea will be measured with a visual analog scale (VAS) and a validated multidimensional dyspnea profile (MDP). The effect of treatment on counterirritation will be measured by recording LEP obtained using a CO2 laser system. The amplitude of the N2-P2 component of the LEP is the main study outcome.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-smoking

Exclusion Criteria:

* acute or chronic pain
* antalgic or psychoactive drugs use
* nefopam hypersensibility
* severe allergy
* diabetes
* glaucoma
* prostate adenoma
* seizure disorder or convulsion history
* heart or circulation disease
* pulmonary disease or asthma
* kidney or liver disease
* brain or nerve disease
* lack of adhesion to no antalgic drug, alcohol, coffee and cola within previous experiment day consumption

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
variation of N2-P2 (components of laser evoked potential - tool of pain measurement)amplitude with inspiratory loading induced by intervention | Change from baseline to 1 hour and half from intervention
  LEP will be recorded before intervention at baseline and after intervention at baseline, during inspiratory loading and recovery. The outcome is the variation of N2-P2 amplitude with inspiratory loading induced by intervention

SECONDARY OUTCOMES:
variation of subject rating of breathing discomfort (dyspnea) | Change from baseline to 1 hour and half from intervention
  repeated measurement on VAS (visual analog scale)
variation of N20-P25 amplitude (components of somesthesic evoked potential (SEP) -measurement of sensitivity) | Change from baseline to 1 hour and half from intervention
  SEP will be recorded before intervention at baseline and after intervention at baseline, during inspiratory loading. This is a methodological control

CONTACTS AND LOCATIONS:
Overall Officials: Capucine Morelot, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Pitié salpetriere Hospital, Paris, France